CLINICAL TRIAL: NCT03517410
Title: Association Between the Duration of Smart Phone Use and Back Dysfunction in Patients With Chronic Mechanical Low Back Pain
Brief Title: Association Between the Duration of Smart Phone Use and Back Dysfunction in Patients With Low Back Pain
Status: Completed | Type: Observational
Sponsor: Aliaa Rehan Youssef (Other)
Responsible Party: Sponsor-Investigator, Aliaa Rehan Youssef, Associate Professor of Orthopedic Physical Therapy, Cairo University
Organization: Cairo University (Other)
Other Study IDs: MWahba
Record Dates: First submitted 2018-04-25; First posted 2018-05-07 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Mechanical Low Back Pain
Keywords: Mechanical Low Back Pain; Smart phone; Low Back Pain; Chronic Mechanical Low Back Pain; CLBP
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smart phone Use Experimental group: Patients with CLBP
  Interventions: Other: Smart phone use

INTERVENTIONS:
Other: Smart phone use — Patients will be asked to use the smart phone while seated for either: (1) 10 minutes or (2) 30 minutes.

SUMMARY:
This study investigates the association between the duration of smart phone use and back pain and proprioception deficits in patients with chronic mechanical low back pain (CLBP).

It is hypothesized that increased duration of smart phone use will be associated with

1. Increased back pain as measured by the Visual Analogue Scale (VAS)
2. Reduced proprioception acuity as indicated by increased angle of error of back repositioning as measured by isokinetic dynamometer.

DETAILED DESCRIPTION:
After patient screening against inclusion and exclusion criteria, eligible patients will be informed about the aim of the study and all testing procedures. Then, they will be asked to participate in the study, if agreed an informed consent will be signed . Basic demographic information as well as questions regarding the average daily smart phone use will be collected .

Patient will be tested in two separate sessions. During each session, the participant will be given a standardized phone and will be asked to play a standardized game "subway surfers " from a standardized sitting position for 10 or 30 minutes.

Pain and back repositioning error will be measured before and after the smart phone use. Pain will be measured first, then repositioning error.

Pain measurement:

Each participant will be instructed to rate the current level of pain by placing a mark across the horizontal VAS line. The distance in millimeters from the lower limit will be measured using a ruler.

Proprioception acuity:

Biodex isokinetic system preparation:

First, the system will be calibrated according to the manufacturer guidelines. For initialization of the Biodex system, the device, computer and dynamometer power will be switched on and all device attachments will be removed. Then, the start key in the control panel will be pressed. Few seconds will be allowed for the dynamometer shaft to rotate freely until the system displays a message that it is initializing the dynamometer. Once the initialization procedure is completed, the start key will be pressed again as indicated by the system status window. The personal data of each subject will be entered into the computer.

Repositioning error measurement:

Each participant will then be seated on the Biodex chair with his or her low back fitted backwards against the lumbar pad. Both knees will be fixed in place using two anterior curved leg pads. Legs will be kept relaxed vertically with both feet off the ground. The upper trunk will be fastened to the back of the chair using a belt. Both thighs will be fastened to the chair using straps while forearms will be kept crossed over the chest. The seat will be adjusted to allow the axis of rotation of the dynamometer to be at the level of L5/S1 disc space. Participants will be instructed to close their eyes during test performance. The limits of available range of motion (ROM) will determined for each participant by starting at the 0° position (neutral sitting with hips flexed 90°) and then instructing the participant to flex his or her trunk as much as possible to determine the available ROM in flexion and examine his or her ability to reach the target position for the isokinetic test (30° of lumbar flexion). The dynamometer will be locked in the 0° position to provide a fixed starting position for all participants during all trials The chosen protocol allows the participants to perform 1 familiarization trial followed by 1 actual test; this step will be repeated 3 times so that there will be 3 familiarization trials and 3 actual testing procedures. The average of the 3 actual testing results will be retrieved from the isokinetic device software. During the familiarization trial and after covering the eyes, participant will be instructed to flex his or her trunk until it is stopped by the machine at 30° of flexion. This position will be held for 5 seconds. The patients will be instructed to remember this position in order to reproduce it as precisely as possible during the subsequent actual test procedure. During the actual test procedure, the tested participants will press a hold button when they assume the target position to allow the device to record and save the reached angle. During the data collection process, no visual (eyes will be closed) or verbal feedback will be provided for the participants.

The results of the test will be recorded and printed by the isokinetic machine. It will include the value of error of every trial and the average error of the 3 trials.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian adult patients with mechanical CLBP Back pain duration is greater than 3 months Age ranging from 18 years to 45

Exclusion Criteria:

* Patients with any systemic disease that may affect spine function.
* Patients with previous history of spine trauma or dysfunction other than mechanical LBP.
* Lumbosacral nerve root entrapment.
* Patients with memory loss or impaired cognitive function
* patients who report back pain associated with sitting position

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Seventy male and female adults will be recruited from out patient clinic of the faculties of Physical therapy and medicine, Cairo University. Further, physical therapy students who are diagnosed with CLBP will be recruited via advertising on social media.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Pain | same day
  Current pain intensity will be measured using the Visual Analogue Scale (VAS). This scale is a 100 mm line drawn on a piece of paper. The line is labeled 0 at one end (indicating no pain) and 10 at the other end (indicating excruciating pain). A change of minimally 20 mm on VAS is considered a minimal detectable change.

SECONDARY OUTCOMES:
Back repositioning error in flexion direction | Same day
  Back repositioning error flexion as measured using Biodex isokinetic system 3 at 30 degree angle flexion

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Rehan Youssef, PhD, Principal Investigator — Cairo University; Dina Othman Shokri, PhD, Study Director — Faculty of Physical Therapy, Badr University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Alhalabi MS, Alhaleeb H, Madani S. Risk factors associated with chronic low back pain in Syria. Avicenna J Med. 2015 Oct-Dec;5(4):110-6. doi: 10.4103/2231-0770.165123. PMID 26629465
- [Background] Ali M, Asim M, Danish SH, Ahmad F, Iqbal A, Hasan SD. Frequency of De Quervain's tenosynovitis and its association with SMS texting. Muscles Ligaments Tendons J. 2014 May 8;4(1):74-8. eCollection 2014 Jan. PMID 24932451
- [Background] Atlas SJ, Deyo RA. Evaluating and managing acute low back pain in the primary care setting. J Gen Intern Med. 2001 Feb;16(2):120-31. doi: 10.1111/j.1525-1497.2001.91141.x. PMID 11251764
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Balakrishnan, R., Chinnavan, E., & Feii, T. (2016). An extensive usage of hand held devices will lead to musculoskeletal disorder of upper extremity among student in AMU : A survey method. International Journal of Physical Education, Sport and Health, 3(2), 368-372.
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Chany AM, Marras WS, Burr DL. The effect of phone design on upper extremity discomfort and muscle fatigue. Hum Factors. 2007 Aug;49(4):602-18. doi: 10.1518/001872007X215683. PMID 17702212
- [Background] Borenstein DG. Chronic low back pain. Rheum Dis Clin North Am. 1996 Aug;22(3):439-56. doi: 10.1016/s0889-857x(05)70281-7. PMID 8844907
- [Background] Chiang HY, Liu CH. Exploration of the associations of touch-screen tablet computer usage and musculoskeletal discomfort. Work. 2016 Mar 10;53(4):917-25. doi: 10.3233/WOR-162274. PMID 26967038
- [Background] Deyo RA. Early diagnostic evaluation of low back pain. J Gen Intern Med. 1986 Sep-Oct;1(5):328-38. doi: 10.1007/BF02596214. No abstract available. PMID 2945917
- [Background] Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis. 1978 Aug;37(4):378-81. doi: 10.1136/ard.37.4.378. PMID 686873
- [Background] Drouin JM, Valovich-mcLeod TC, Shultz SJ, Gansneder BM, Perrin DH. Reliability and validity of the Biodex system 3 pro isokinetic dynamometer velocity, torque and position measurements. Eur J Appl Physiol. 2004 Jan;91(1):22-9. doi: 10.1007/s00421-003-0933-0. Epub 2003 Sep 24. PMID 14508689
- [Background] Garcia-Vaquero MP, Barbado D, Juan-Recio C, Lopez-Valenciano A, Vera-Garcia FJ. Isokinetic trunk flexion-extension protocol to assess trunk muscle strength and endurance: Reliability, learning effect, and sex differences. J Sport Health Sci. 2020 Dec;9(6):692-701. doi: 10.1016/j.jshs.2016.08.011. Epub 2016 Nov 14. PMID 33308821
- [Background] Georgy EE. Lumbar repositioning accuracy as a measure of proprioception in patients with back dysfunction and healthy controls. Asian Spine J. 2011 Dec;5(4):201-7. doi: 10.4184/asj.2011.5.4.201. Epub 2011 Nov 28. PMID 22164313
- [Background] Gustafsson E, Johnson PW, Lindegard A, Hagberg M. Technique, muscle activity and kinematic differences in young adults texting on mobile phones. Ergonomics. 2011 May;54(5):477-87. doi: 10.1080/00140139.2011.568634. PMID 21547792
- [Background] Haug S, Castro RP, Kwon M, Filler A, Kowatsch T, Schaub MP. Smartphone use and smartphone addiction among young people in Switzerland. J Behav Addict. 2015 Dec;4(4):299-307. doi: 10.1556/2006.4.2015.037. PMID 26690625
- [Background] Heikkila HV, Wenngren BI. Cervicocephalic kinesthetic sensibility, active range of cervical motion, and oculomotor function in patients with whiplash injury. Arch Phys Med Rehabil. 1998 Sep;79(9):1089-94. doi: 10.1016/s0003-9993(98)90176-9. PMID 9749689
- [Background] Hussien HM, Abdel-Raoof NA, Kattabei OM, Ahmed HH. Effect of Mulligan Concept Lumbar SNAG on Chronic Nonspecific Low Back Pain. J Chiropr Med. 2017 Jun;16(2):94-102. doi: 10.1016/j.jcm.2017.01.003. Epub 2017 Mar 30. PMID 28559749
- [Background] Katz JN. Lumbar disc disorders and low-back pain: socioeconomic factors and consequences. J Bone Joint Surg Am. 2006 Apr;88 Suppl 2:21-4. doi: 10.2106/JBJS.E.01273. PMID 16595438
- [Background] Kim SY, Koo SJ. Effect of duration of smartphone use on muscle fatigue and pain caused by forward head posture in adults. J Phys Ther Sci. 2016 Jun;28(6):1669-72. doi: 10.1589/jpts.28.1669. Epub 2016 Jun 28. PMID 27390391
- [Background] Kwon M, Kim DJ, Cho H, Yang S. The smartphone addiction scale: development and validation of a short version for adolescents. PLoS One. 2013 Dec 31;8(12):e83558. doi: 10.1371/journal.pone.0083558. eCollection 2013. PMID 24391787
- [Background] Lee J, Seo K. The comparison of cervical repositioning errors according to smartphone addiction grades. J Phys Ther Sci. 2014 Apr;26(4):595-8. doi: 10.1589/jpts.26.595. Epub 2014 Apr 23. PMID 24764641
- [Background] Lee S, Kang H, Shin G. Head flexion angle while using a smartphone. Ergonomics. 2015;58(2):220-6. doi: 10.1080/00140139.2014.967311. Epub 2014 Oct 17. PMID 25323467
- [Background] Leinonen V, Kankaanpaa M, Luukkonen M, Hanninen O, Airaksinen O, Taimela S. Disc herniation-related back pain impairs feed-forward control of paraspinal muscles. Spine (Phila Pa 1976). 2001 Aug 15;26(16):E367-72. doi: 10.1097/00007632-200108150-00014. PMID 11493866
- [Background] Mayer T, Gatchel R, Betancur J, Bovasso E. Trunk muscle endurance measurement. Isometric contrasted to isokinetic testing in normal subjects. Spine (Phila Pa 1976). 1995 Apr 15;20(8):920-6; discussion 926-7. PMID 7644957
- [Background] Melloh M, Roder C, Elfering A, Theis JC, Muller U, Staub LP, Aghayev E, Zweig T, Barz T, Kohlmann T, Wieser S, Juni P, Zwahlen M. Differences across health care systems in outcome and cost-utility of surgical and conservative treatment of chronic low back pain: a study protocol. BMC Musculoskelet Disord. 2008 Jun 6;9:81. doi: 10.1186/1471-2474-9-81. PMID 18534034
- [Background] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Background] Ming Z, Pietikainen S, Hanninen O. Excessive texting in pathophysiology of first carpometacarpal joint arthritis. Pathophysiology. 2006 Dec;13(4):269-70. doi: 10.1016/j.pathophys.2006.09.001. Epub 2006 Oct 17. PMID 17049823
- [Background] O'Sullivan PB, Burnett A, Floyd AN, Gadsdon K, Logiudice J, Miller D, Quirke H. Lumbar repositioning deficit in a specific low back pain population. Spine (Phila Pa 1976). 2003 May 15;28(10):1074-9. doi: 10.1097/01.BRS.0000061990.56113.6F. PMID 12768152
- [Background] Olaogun, M. O. B., Adedoyin, R. A., Ikem, I. C., & Anifaloba, O. R. (2004). Reliability of rating low back pain with a visual analogue scale and a semantic differential scale. Physiotherapy Theory and Practice, 20(2), 135-142.
- [Background] Ostelo RW, de Vet HC. Clinically important outcomes in low back pain. Best Pract Res Clin Rheumatol. 2005 Aug;19(4):593-607. doi: 10.1016/j.berh.2005.03.003. PMID 15949778
- [Background] Parasuraman S, Sam AT, Yee SWK, Chuon BLC, Ren LY. Smartphone usage and increased risk of mobile phone addiction: A concurrent study. Int J Pharm Investig. 2017 Jul-Sep;7(3):125-131. doi: 10.4103/jphi.JPHI_56_17. PMID 29184824
- [Background] Richter HO, Zetterberg C, Forsman M. Trapezius muscle activity increases during near work activity regardless of accommodation/vergence demand level. Eur J Appl Physiol. 2015 Jul;115(7):1501-12. doi: 10.1007/s00421-015-3125-9. Epub 2015 Feb 20. PMID 25697148
- [Background] Salaffi F, Stancati A, Silvestri CA, Ciapetti A, Grassi W. Minimal clinically important changes in chronic musculoskeletal pain intensity measured on a numerical rating scale. Eur J Pain. 2004 Aug;8(4):283-91. doi: 10.1016/j.ejpain.2003.09.004. PMID 15207508
- [Background] Samaha, M., & Hawi, N. S. (2016). Relationships among smartphone addiction , stress , academic performance , and satisfaction with life. Computers in Human Behavior, 57, 321-325.
- [Background] Shan Z, Deng G, Li J, Li Y, Zhang Y, Zhao Q. Correlational analysis of neck/shoulder pain and low back pain with the use of digital products, physical activity and psychological status among adolescents in Shanghai. PLoS One. 2013 Oct 11;8(10):e78109. doi: 10.1371/journal.pone.0078109. eCollection 2013. PMID 24147114
- [Background] Silva GR, Pitangui AC, Xavier MK, Correia-Junior MA, De Araujo RC. Prevalence of musculoskeletal pain in adolescents and association with computer and videogame use. J Pediatr (Rio J). 2016 Mar-Apr;92(2):188-96. doi: 10.1016/j.jped.2015.06.006. Epub 2015 Dec 28. PMID 26738891
- [Background] O'Sullivan P. Diagnosis and classification of chronic low back pain disorders: maladaptive movement and motor control impairments as underlying mechanism. Man Ther. 2005 Nov;10(4):242-55. doi: 10.1016/j.math.2005.07.001. Epub 2005 Sep 9. PMID 16154380
- [Background] Swinkels A, Dolan P. Regional assessment of joint position sense in the spine. Spine (Phila Pa 1976). 1998 Mar 1;23(5):590-7. doi: 10.1097/00007632-199803010-00012. PMID 9530791
- [Background] Takala EP, Korhonen I, Viikari-Juntura E. Postural sway and stepping response among working population: reproducibility, long-term stability, and associations with symptoms of the low back. Clin Biomech (Bristol). 1997 Oct;12(7-8):429-437. doi: 10.1016/s0268-0033(97)00033-8. PMID 11415752
- [Background] Wilson SE, Granata KP. Reposition sense of lumbar curvature with flexed and asymmetric lifting postures. Spine (Phila Pa 1976). 2003 Mar 1;28(5):513-8. doi: 10.1097/01.BRS.0000048674.75474.C4. PMID 12616167
- [Background] Yoon JO; BHSc; Kang MH, Kim JS; BHSc; Oh JS. The effects of gait with use of smartphone on repositioning error and curvature of the lumbar spine. J Phys Ther Sci. 2015 Aug;27(8):2507-8. doi: 10.1589/jpts.27.2507. Epub 2015 Aug 21. PMID 26357430
- [Background] Oxford Dictionary of English